CLINICAL TRIAL: NCT06811922
Title: Primary Prevention of Intimate Partner Violence
Brief Title: The Primary Prevention of Intimate Partner Violence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ameeta Kalokhe, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007022; 1R01HD114862-01 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Intimate Partner Violence
MeSH Terms: interventions — 1,4-alpha-Glucan Branching Enzyme; Methods

STUDY DESIGN:
Intervention Model Description: Eligible dyads will be sequentially enrolled and randomly assigned within each geographic strata (slum community) of Mumbai and Pune (equal numbers in both cities) using a computer-generated randomization scheme to the GBE intervention (n=500 dyads) or control arm (n=350 dyads); total n=1,700 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GBE (Ghya Bharaari Ekatra) Group (Experimental): * Dyads assigned to the GBE arm will be sequentially assigned into a group composed of 5 newly married (married ≤ 1 yr) couples.
  * GBE will be delivered to groups of 5 newly married couples (husband-wife dyads) in weekly 2-hour sessions over a 6-week period, plus ethical standard of care (information about IPV resources).
  * GBE will be facilitated by a male/female pair of trained peer educators and held at a community-based venue, in the slum communities in which the couples reside.
  * The intervention is highly participatory.
  Interventions: Behavioral: GBE (Ghya Bharaari Ekatra) intervention; Behavioral: Ethical standard of care
- Control Group (Active Comparator): Control groups will solely receive the ethical standard of care (information about IPV resources).
  Interventions: Behavioral: Ethical standard of care

INTERVENTIONS:
Behavioral: GBE (Ghya Bharaari Ekatra) intervention — Ghya Bharaari Ekatra (Marathi for "Take a flight together") intervention
  The intervention consists of six sessions. Each session will cover one of 6 major modules to enhance transformation of motivation: 1) You, Me, and Us: Spending Meaningful Time Together, 2) I'm a Champion: I Can't Be Broken and I don't Accept Defeat! 3) Building Communication and conflict management strategies, and 4) Empowerment of the Couple: Planning Ahead, 5) Sexual communication and the sexual relationships, and 6) A Lens into Domestic Violence. The sessions will be audio-recorded and include a combination of didactics, interactive discussions, media use, and role play. The expected durations of sessions are 2 hours.
  GBE will be delivered to a total of 500 dyads.
  Other Names: Ghya Bharaari Ekatra intervention; Take a flight together intervention; IPV Intervention
  Arms: GBE (Ghya Bharaari Ekatra) Group
Behavioral: Ethical standard of care — Ethical standard of care includes information on IPV and mental and reproductive/sexual health resources) to prevent IPV experience. This intervention will be delivered to a total of 350 dyads.

SUMMARY:
This is a cluster randomized trial for newly married dyads, that seeks to quantify the impact of GBE's (Ghya Bharaari Ekatra's) intervention on intimate partner violence (IPV) and downstream outcomes, mental health and reproductive autonomy, examine its mechanism of action, contexts in which it may need modification, and factors associated with its future successful adoption and implementation.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) is experienced by one-fourth of women in India and associated with poor mental, physical, sexual and reproductive health, leading many experts including the World Health Organization to call for the urgent development of effective primary IPV prevention. The investigators previously developed an evidence-based, theory-driven, dyadic intervention, Ghya Bharaari Ekatra (GBE, "Take a Flight Together," NIH/FIC K01 TW009664) for the primary prevention of IPV among newly married couples residing in slums in India. GBE is delivered over six weekly sessions by a team of lay peer educators to groups of five couples and makes use of engaging culturally tailored delivery methods to challenge norms and build knowledge and skills to address six key IPV determinants: limited relationship quality time, poor self-esteem, resilience, communication and conflict management, sexual communication and sexual/reproductive health knowledge, and conservative IPV norms and definitions. In a pilot study of 40 couples married < 1 year, it was found that GBE demonstrated high acceptance (with 85% of participants retained across all 6 sessions), feasibility, safety (no reported adverse events), and preliminary efficacy in preventing IPV and improving mental health in the female partner. The investigators now seek to quantify GBE's impact on IPV and downstream outcomes, mental health and reproductive autonomy, examine its mechanism of action, contexts in which it may need modification, and factors associated with its future successful adoption and implementation.

The research team hypothesizes that (1) GBE prevents IPV experience and enhances reproductive autonomy among women,(2) GBE improves mental health among both dyadic members, and (3) GBE's effects are mediated by the IPV determinants it was designed to address. The team, with 15 years of IPV research experience in India, proposes a cluster randomized trial of 850 newly married dyads (500 to GBE and 350 controls) in Maharashtra, India to execute the following aims: 1) to quantify the impact of the GBE intervention compared to the ethical standard of care (information on IPV and mental and reproductive/sexual health resources) in preventing IPV experience (primary outcome), enhancing reproductive autonomy among newly married women (secondary outcome) and mental health among the both members of the dyad (secondary outcome) at 12 months; 2) to conduct mediation and moderation analyses for the efficacy of the GBE intervention; and 3) to identify barriers, facilitators, and strategies for future, successful adoption and implementation of GBE through exit interviews with GBE participants and qualitative interviews, guided by Consolidated Framework for Implementation Research, with interventionists, adopters, and other stakeholders who have influence over implementation outcomes. Study findings will provide the information necessary to facilitate scale-up of GBE across India and similar resource-limited, high-burden settings globally upon study completion.

ELIGIBILITY:
Inclusion Criteria:

* couples wherein both members are age ≥18 years,
* married ≤ 1 year, in their first marriage, married to only one individual, cohabiting in a slum in Mumbai or Pune India, and
* fluent in Marathi and/or Hindi
* Both members of the couple must meet eligibility criteria and be present at the session for the couple to participate.

Exclusion Criteria:

* As GBE was designed for primary IPV prevention, couples in which the female member screens positive for physical and/or sexual IPV (using the modified Conflict Tactics Scale (CTS-2)) at baseline will be excluded (and referred to support services)
* those in the 3rd trimester of pregnancy (as women traditionally return to their natal home during this perinatal period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Intimate Partner Violence (IPV) Experience | 12 months post intervention
  IPV experience is defined as a woman experiencing one or more act of physical, sexual, and/or psychological IPV.

SECONDARY OUTCOMES:
Change in General Health Questionnaire-12 (GHQ-12) Score | Baseline, 6 and 12 months post intervention
  Mental health is assessed using the General Health Questionnaire-12 (GHQ-12). The GHQ-12 is scored using a 4-point Likert scale, where each item is assigned a value from 0 to 3, resulting in a total score ranging from 0 to 36, with higher scores indicating greater psychological distress.
Change in Reproductive Autonomy Scale (RAS) Score | Baseline, 6 and 12 months post intervention
  Reproductive autonomy among women is measured using a culturally-tailored version of the Reproductive Autonomy Scale (RAS). The RAS is a 14-item self-reported measure of individual experiences of ability to achieve reproductive goals, comprising of three domains: Decision-making, Freedom from Coercion, and Communication. The Decision-making subscale uses a 3-point Likert scale, where each item is assigned a value of 1 to 3. The Freedom from Coercion and Communication Subscales use a 4-point Likert scale, where each item is assigned a value of 1 to 4. Item scores are averaged to calculate subscale and total measure scores. Higher scores indicate greater levels of autonomy.

CONTACTS AND LOCATIONS:
Overall Officials: Ameeta Kalokhe, MD, Principal Investigator — Emory University
Locations (2):
- India (2):
  - Indian Council of Medical Research-National Institute for Research in Reproductive and Child Health (ICMR-NIRRCH),, Mumbai, Maharashtra
  - Indian Council of Medical Research - National Institute of Translational Virology and AIDS Research (ICMR-NITVAR), Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: Yes
Individual participant survey data collected during the trial that underlie the results reported, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made as soon as possible, and no later than the time of publication, or end of the funding period, whichever comes first. Data will remain available indefinitely.
Access Criteria: Globally available to researchers from academic institutions for intervention, program, or policy development. Restrictions will be outlined in the Restricted Data Use Agreement.
  Data will be available to achieve aims in an approved proposal. Data will be deposited in Data Sharing Demographic Research (DSDR). Must be using a secure server to access data. To gain access, data requestors must ensure request conforms to restrictions outlined in the Restricted Use Data Agreement.